CLINICAL TRIAL: NCT05887544
Title: Towards Objective Dietary Assessment in Large-scale Studies
Acronym: ODA
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M244
Record Dates: First submitted 2023-04-25; First posted 2023-06-02 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: sampling; food intake biomarkers; type 2 diabetes; urine; blood; hair; diet assessment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Yogurt; Food

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine and hair samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes: Overall study population. In addition, a subset of volunteer participants (up to 20 participants) will be asked to consume extra portions of fermented dairy products (skyr, ymer and yogurt) 1-2 days before the spot urine sample to be able to validate markers for specific foods.
  Interventions: Other: Exposure: Plant-based diet pattern; Other: Intervention: Fermented dairy products; Other: Exposure: individual foods and food groups

INTERVENTIONS:
Other: Exposure: Plant-based diet pattern — From dietary records average intake across food groups will be calculated and a plant-based diet index score will be generated to group participants.
  Other Names: Plant-based diet index
Other: Intervention: Fermented dairy products — 1000g of the product to be consumed 1-2 days prior to spot urine sample.
  Other Names: Commercially available skyr, ymer and yogurt
Other: Exposure: individual foods and food groups — From the dietary records, average intake of specific foods or food groups will be calcualted.
  Other Names: Foods and food groups

SUMMARY:
Enabling an objective measure of diet, covering individual foods as well as different dietary patterns, in large-scale studies has great potential; this would for instance improve our understanding of the role of diet in long-term disease prevention and care in people with type 2 diabetes.

The overarching aim of this study is to develop a framework from which dietary intake can be assessed, both as single foods and dietary patterns, in cohort studies among people with type 2 diabetes. This study is performed to assess which collection strategy best reflects long-term dietary intake and to weigh this up against feasibility and costs in large-scale studies.

DETAILED DESCRIPTION:
This is a 4-week observational study that will be carried out in adults with newly diagnosed type 2 diabetes living in Denmark.

The aim is to recruit up to 60 participants aged 18-75. The participants will be asked to record and weight their habitual food intake on 8 days spread out within a one-month time period. They will also be asked to complete one 24-hour urine collection the day before study start and provide 7 morning spot urine samples on the subsequent mornings after filling in the food diary.

At the start of the study period participants will undergo a DXA scan and have a blood sample taken. At the end of the study period a second blood sample will be drawn and a hair sample will also be collected. Incomplete 24-hour collections will be judged based on predicted 24-hour creatinine excretion from lean body mass and actual creatinine excretion being in the interval from 0.8-1.2, which corresponds to ~20% on each side of the expected excretion. Participants falling outside this interval will be asked to complete a new 24-hour urine sample. As the primary aim of this study is validation, it is important that the samples provided are as complete as possible.

In the one-month period between visits to the study center, a subset of volunteer participants (up to 20 participants) will be asked to consume extra portions of fermented dairy products (skyr, ymer and yogurt) 1-2 days before the spot urine sample to be able to validate markers for specific foods. All participants in the subcohort will consume each of the foods one time before a spot urine and one time be asked to abstain intake of dairy products as a control. Foods will be provided to the participants.

Note: the study has ended with fewer participants than expected due to problems with recruitment. We will analyse these samples and work on samples from another study to answer our initial research questions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes (within the last 5 years from study start) (self-reported)
* 18.5-35.0 kg/m2 BMI
* More than 1cm of natural hair on the head
* Have not dyed their hair in the previous 6 months
* Willing to record dietary intake up to 9 days
* Willing to have blood samples drawn two times
* Willing to collect up to two 24-hour urine samples and 7 spot urine samples at home and be able to store them in their own freezer in provided tubes and boxes throughout the one-month study
* Have no intention to radically change dietary and physical activity habits during the study period
* Owning a smartphone with internet connection
* Can speak and read Danish

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosed with any chronic or communicable diseases including liver diseases (e.g., active hepatitis B and C infections), liver cirrhosis, severe psychiatric illness or any other clinical condition that makes the subject ineligible according to the clinically responsible medical doctor (except type 2 diabetes) (self-reported).
* History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
* Diagnosed with any CVD event (e.g., myocardial infarction, revascularization procedure or stroke) within the past 2 years
* Unintentional weight loss >20% during the last 6 months
* Regular intake of prescription medication (except diabetes medication, blood pressure-lowering medication, cholesterol-lowering medication, mild antidepressants or contraceptive pills)
* Concurrent participation in another trial
* Not willing to sign the Informed consent form (ICF)
* Not willing to comply with the all the trial procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with newly diagnosed type 2 diabetes that are otherwise generally health and willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Concentration of Indole-3-lactic acid in blood | 1 month
  Difference in beta-coefficient of the concentration of Indole-3-lactic acid (https://hmdb.ca/metabolites/HMDB0000671) in blood measured at the end of the study between those consuming fermented dairy products compared to participants not consuming fermented dairy products. A linear regression model will be used with Indole-3-lactic acid concentration as the outcome and consuming vs not consuming fermented dairy products as the exposure.
  Indole-3-lactic acid in blood will be analysed using an ultra-performance liquid chromatography (UPLC) system coupled to a quadrupole time-of-flight mass spectrometer (ViON QTOF, Waters Corporation, Manchester, UK).

SECONDARY OUTCOMES:
Concentration of Indole-3-lactic acid in urine | 1 month
  Difference in beta-coefficient of the concentration of Indole-3-lactic acid (https://hmdb.ca/metabolites/HMDB0000671) in the average of 7 spot urine samples between those consuming fermented dairy products compared to participants not consuming fermented dairy products. A linear regression model will be used with Indole-3-lactic acid concentration as the outcome and consuming vs not consuming fermented dairy products as the exposure.
  Indole-3-lactic acid in urine will be analysed using an ultra-performance liquid chromatography (UPLC) system coupled to a quadrupole time-of-flight mass spectrometer (ViON QTOF, Waters Corporation, Manchester, UK).
Concentration of 3-Phenyllactic acid in blood | 1 month
  Difference in beta-coefficient of the concentration of 3-Phenyllactic acid (https://hmdb.ca/metabolites/HMDB0000779) in blood measured at the end of the study between those consuming fermented dairy products compared to participants not consuming fermented dairy products. A linear regression model will be used with 3-Phenyllactic acid concentration as the outcome and consuming vs not consuming fermented dairy products as the exposure.
  Indole-3-lactic acid in blood will be analysed using an ultra-performance liquid chromatography (UPLC) system coupled to a quadrupole time-of-flight mass spectrometer (ViON QTOF, Waters Corporation, Manchester, UK).
Concentration of 3-Phenyllactic acid in urine | 1 month
  Difference in beta-coefficient of the concentration of 3-Phenyllactic acid (https://hmdb.ca/metabolites/HMDB0000779) in the average of 7 spot urine samples between those consuming fermented dairy products compared to participants not consuming fermented dairy products. A linear regression model will be used with 3-Phenyllactic acid concentration as the outcome and consuming vs not consuming fermented dairy products as the exposure.
  Indole-3-lactic acid in urine will be analysed using an ultra-performance liquid chromatography (UPLC) system coupled to a quadrupole time-of-flight mass spectrometer (ViON QTOF, Waters Corporation, Manchester, UK).

OTHER OUTCOMES:
Exploratory analyses | 1 day or 1 month
  Metabolite signatures of a plant-based dietary pattern from one morning spot urine vs average of 7 morning spot urine samples. The study will investigate whether the classification of participants into groups of adherence to a plant-based diet is significantly more accurate for a metabolite signature of a plant-based diet based on the average of 7 morning spot urine samples than for a metabolite signature based on a single morning spot urine sample.
  A similar approach will be used to:
  * Compare the blood (serum) sample at study start with the 7 spot urine samples
  * Compare food intake biomarkers from the 24-hour urine samples with a single spot urine sample using the 1 day food diary completed on the same day as reference for true intake
  * Compare food intake biomarkers from a single spot urine sample with a blood sample, both from the start or end of the study
  * Compare metabolites from blood samples at study start with blood samples at end of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Once the project is finished, data will by fully anonymised and shared with other researchers.
Supporting Information: Study Protocol
Time Frame: After completion of the main study project.
Access Criteria: Will be uploaded on University of Copenhagen data sharing platform. More information to come.